CLINICAL TRIAL: NCT03369223
Title: A Phase 1/2 First-in-Human Study of BMS-986249 Alone and in Combination With Nivolumab in Advanced Solid Tumors
Brief Title: A Study of BMS-986249 Alone and in Combination With Nivolumab in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA030-001; 2018-000416-21 (EudraCT Number)
Record Dates: First submitted 2017-12-06; First posted 2017-12-11 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Advanced Cancer
Keywords: Antibodies; Antineoplastic Agents; Immunologic Factors; Nivolumab; Antibodies, Monoclonal; Physiological Effects of Drugs
MeSH Terms: interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part 1A: BMS-986249 (Experimental)
  Interventions: Biological: BMS-986249
- Part 1B: BMS-986249 + nivolumab (nivo) (Experimental)
  Interventions: Biological: BMS-986249; Biological: Nivolumab
- Part 2A Arm C: BMS-986249 + nivo (Experimental): Previously untreated unresectable stage III-IV melanoma
  Interventions: Biological: BMS-986249; Biological: Nivolumab
- Part 2A Arm D: ipilimumab + nivo then nivo (Experimental): Previously untreated unresectable stage III-IV melanoma
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Part 2A Arm F: BMS-986249 + nivo (Experimental): Previously untreated unresectable stage III-IV melanoma
  Interventions: Biological: BMS-986249; Biological: Nivolumab
- Part 2B Cohort 1: BMS-986249 + nivo (Experimental): Advanced or intermediate hepatocellular carcinoma (HCC)
  Interventions: Biological: BMS-986249; Biological: Nivolumab
- Part 2B Cohort 2: BMS-986249 + nivo (Experimental): Metastatic castration-resistant prostate cancer (CRPC)
  Interventions: Biological: BMS-986249; Biological: Nivolumab
- Part 2B Cohort 3: BMS-986249 + nivo (Experimental): Unresectable locally advanced or metastatic triple-negative breast cancer (TNBC)
  Interventions: Biological: BMS-986249; Biological: Nivolumab
- Part 2A Arm A: BMS-986249 + nivo then nivo (Experimental): * Previously untreated unresectable stage III-IV melanoma
  * Enrollment is closed for this Arm
  Interventions: Biological: BMS-986249; Biological: Nivolumab
- Part 2A Arm B: BMS-986249 + nivo (Experimental): * Previously untreated unresectable stage III-IV melanoma
  * Enrollment is closed for this Arm
  Interventions: Biological: BMS-986249; Biological: Nivolumab
- Part 2A Arm E: Nivo (Experimental): * Previously untreated unresectable stage III-IV melanoma
  * Enrollment is closed for this Arm
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: BMS-986249 — Specified dose on specified days
  Arms: Part 1A: BMS-986249; Part 1B: BMS-986249 + nivolumab (nivo); Part 2A Arm A: BMS-986249 + nivo then nivo; Part 2A Arm B: BMS-986249 + nivo; Part 2A Arm C: BMS-986249 + nivo; Part 2A Arm F: BMS-986249 + nivo; Part 2B Cohort 1: BMS-986249 + nivo; Part 2B Cohort 2: BMS-986249 + nivo; Part 2B Cohort 3: BMS-986249 + nivo
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
  Arms: Part 1B: BMS-986249 + nivolumab (nivo); Part 2A Arm A: BMS-986249 + nivo then nivo; Part 2A Arm B: BMS-986249 + nivo; Part 2A Arm C: BMS-986249 + nivo; Part 2A Arm D: ipilimumab + nivo then nivo; Part 2A Arm E: Nivo; Part 2A Arm F: BMS-986249 + nivo; Part 2B Cohort 1: BMS-986249 + nivo; Part 2B Cohort 2: BMS-986249 + nivo; Part 2B Cohort 3: BMS-986249 + nivo
Biological: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy; BMS-734016
  Arms: Part 2A Arm D: ipilimumab + nivo then nivo

SUMMARY:
The purpose of this study is to determine whether BMS-986249 both by itself and in combination with Nivolumab is safe and tolerable in the treatment of advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of a solid tumor that is advanced (metastatic, recurrent, and/or unresectable) with measurable disease or metastatic disease documented by either bone lesions on radionuclide bone scan and/or soft tissue lesions on CT/MRI for prostate cancer and have at least 1 lesion accessible for biopsy. For Part 2B participants with HCC, intermediate disease is allowed.
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Must have received, and then progressed, relapsed, or been intolerant to, at least 1 standard treatment regimen in the advanced or metastatic setting according to tumor type, if such a therapy exists
* Prior anti-cancer treatments such as chemotherapy, radiotherapy, or hormonal are permitted for some participants
* Willing and able to comply with all study procedures

Exclusion Criteria:

* Primary central nervous system (CNS) malignancies, tumors with CNS metastases as the only site of disease or active brain metastases will be excluded
* Other active malignancy requiring concurrent intervention
* Prior organ allograft
* Active, known, or suspected autoimmune disease

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (45):
- United States (19):
  - Local Institution - 0005, Aurora, Colorado
  - Local Institution - 0006, Denver, Colorado
  - Local Institution - 0017, Miami, Florida
  - Local Institution - 0024, Baltimore, Maryland
  - Local Institution - 0001, Hackensack, New Jersey
  - Local Institution - 0002, New York, New York
  - Local Institution - 0003, New York, New York
  - Local Institution - 0029, Cincinnati, Ohio
  - Local Institution - 0013, Eugene, Oregon
  - Local Institution - 0004, Philadelphia, Pennsylvania
  - Local Institution - 0008, Greenville, South Carolina
  - Local Institution - 0010, Austin, Texas
  - Local Institution - 0009, Dallas, Texas
  - Local Institution - 0021, Houston, Texas
  - Local Institution - 0016, San Antonio, Texas
  - Local Institution - 0011, Tyler, Texas
  - Local Institution - 0012, Leesburg, Virginia
  - Local Institution - 0007, Norfolk, Virginia
  - Local Institution - 0018, Vancouver, Washington
- Argentina (3):
  - Local Institution - 0038, Buenos Aires, Distrito Federal
  - Local Institution - 0052, CABA, Distrito Federal
  - Local Institution - 0037, Buenos Aires
- Australia (4):
  - Local Institution - 0015, North Sydney, New South Wales
  - Local Institution - 0014, Adelaide, South Australia
  - Local Institution - 0025, Frankston, Victoria
  - Local Institution - 0047, Heidelberg, Victoria
- Canada (2):
  - Local Institution - 0026, Edmonton, Alberta
  - Local Institution - 0056, Ottawa, Ontario
- Local Institution - 0036, Santiago, Santiago Metropolitan, Chile
- Local Institution - 0039, Helsinki, Finland
- Germany (3):
  - Local Institution - 0030, Essen
  - Local Institution - 0035, Hamburg
  - Local Institution - 0031, Heidelberg
- Italy (3):
  - Local Institution - 0048, Milan
  - Local Institution - 0020, Napoli
  - Local Institution - 0049, Siena
- Local Institution - 0040, Warsaw, Poland
- Romania (2):
  - Local Institution - 0045, Bucharest
  - Local Institution - 0041, Craiova
- Spain (6):
  - Local Institution - 0042, Badalona, Barcelona [Barcelona]
  - Local Institution - 0022, Madrid, Madrid, Comunidad de
  - Local Institution - 0044, Barcelona
  - Local Institution - 0023, Madrid
  - Local Institution - 0050, Madrid
  - Local Institution - 0043, Málaga

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1A: BMS-986249 240 mg Monotherapy: BMS-986249 240 mg IV every 4 weeks (Q4W), up to 2 years
- Part 1A: BMS-986249 800 mg Monotherapy: BMS-986249 800 mg IV every 4 weeks (Q4W), up to 2 years
- Part 1A: BMS-986249 1600 mg Monotherapy: BMS-986249 1600 mg IV every 4 weeks (Q4W), up to 2 years
- Part 1A: BMS-986249 2400 mg Monotherapy: BMS-986249 2400 mg IV every 4 weeks (Q4W), up to 2 years
- Part 1A: BMS-986249 1600 mg Q8W Monotherapy: BMS-986249 1600 mg IV every 8 weeks (Q8W), up to 2 years
- Part 1B: BMS-986249 240 mg Q4W + Nivolumab Combination: BMS-986249 240 mg IV every 4 weeks (Q4W) + nivolumab 480 mg IV Q4W, up to 2 years
- Part 1B: BMS-986249 800 mg Q4W+ Nivolumab Combination: BMS-986249 800 mg IV every 4 weeks (Q4W) + nivolumab 480 mg IV Q4W, up to 2 years
- Part 1B: BMS-986249 1200 mg Q4W + Nivolumab Combination: BMS-986249 1200 mg IV every 4 weeks (Q4W) + nivolumab 480 mg IV Q4W, up to 2 years
- Part 1B: BMS-986249 800 mg Q8W + Nivolumab Combination; Part 2A: Melanoma Arm B: BMS-986249 800 mg + Nivolumab 480 mg Q4W: BMS-986249 800 mg IV every 8 weeks (Q8W) + nivolumab 480 mg IV every 4 weeks (Q4W), up to 2 years
- Part 1B: BMS-986249 1200 mg Q8W+ Nivolumab Combination; Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W; Part 2B: Cohort 1 (Advanced or Intermediate HCC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg IV Q4W; Part 2B: Cohort 2 (Metastatic CRPC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W; Part 2B: Cohort 3 (Unresectable TNBC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W: BMS-986249 1200 mg IV every 8 weeks (Q8W) + nivolumab 480 mg IV every 4 weeks (Q4W), up to 2 years
- Part 1B: BMS-986249 1600 mg Q8W+ Nivolumab Combination: BMS-986249 1600 mg IV every 8 weeks (Q8W) + nivolumab 480 mg IV every 4 weeks (Q4W), up to 2 years
- Part 2A: Melanoma Arm A: BMS-986249 240 mg Q3W + Nivolumab 360 mg Q3W: BMS-986249 240 mg IV every 3 weeks (Q3W) + nivolumab 360 mg IV every 3 weeks (Q3W) (4 doses), then nivolumab 480 mg IV every 4 weeks (Q4W) (maintenance), up to 2 years.
- Part 2A: Melanoma Arm D: Ipilimumab 3 mg/kg Q3W + Nivolumab 1 mg/kg Q3W: Ipilimumab 3 mg/kg IV every 3 weeks (Q3W) + nivolumab 1 mg/kg IV Q3W (4 doses), then nivolumab 480 mg IV every 4 weeks (Q4W) monotherapy, up to 2 years.
- Part 2A: Melanoma Arm E: Nivolumab 480 mg Q4W Monotherapy: Nivolumab 480 mg IV every 4 weeks (Q4W) monotherapy, up to 2 years.
- Part 2A: Melanoma Arm F: BMS-986249 600 mg Q4W + Nivolumab 480 mg Q4W: BMS-986249 600 mg IV every 4 weeks (Q4W) + nivolumab 480 mg IV Q4W, up to 2 years.
Period: Overall Study
Arm/Group | Part 1A: BMS-986249 240 mg Monotherapy | Part 1A: BMS-986249 800 mg Monotherapy | Part 1A: BMS-986249 1600 mg Monotherapy | Part 1A: BMS-986249 2400 mg Monotherapy | Part 1A: BMS-986249 1600 mg Q8W Monotherapy | Part 1B: BMS-986249 240 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q4W+ Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q8W + Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q8W+ Nivolumab Combination | Part 1B: BMS-986249 1600 mg Q8W+ Nivolumab Combination | Part 2A: Melanoma Arm A: BMS-986249 240 mg Q3W + Nivolumab 360 mg Q3W | Part 2A: Melanoma Arm B: BMS-986249 800 mg + Nivolumab 480 mg Q4W | Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2A: Melanoma Arm D: Ipilimumab 3 mg/kg Q3W + Nivolumab 1 mg/kg Q3W | Part 2A: Melanoma Arm E: Nivolumab 480 mg Q4W Monotherapy | Part 2A: Melanoma Arm F: BMS-986249 600 mg Q4W + Nivolumab 480 mg Q4W | Part 2B: Cohort 1 (Advanced or Intermediate HCC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg IV Q4W | Part 2B: Cohort 2 (Metastatic CRPC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2B: Cohort 3 (Unresectable TNBC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W
Started (Started= Directly Treated Part 1 A and B, or randomized Part 2A and 2 B) | 6 | 11 | 10 | 1 | 11 | 12 | 11 | 9 | 13 | 9 | 10 | 3 | 3 | 58 | 59 | 3 | 36 | 5 | 41 | 45
Treated | 6 | 11 | 10 | 1 | 11 | 12 | 11 | 9 | 13 | 9 | 10 | 3 | 3 | 57 | 58 | 3 | 36 | 5 | 41 | 45
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 6 | 7 | 1 | 2 | 0 | 1 | 3
Not Completed | 6 | 11 | 10 | 1 | 11 | 12 | 11 | 9 | 13 | 8 | 10 | 3 | 3 | 52 | 52 | 2 | 34 | 5 | 40 | 42
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Participant no longer meets study criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Not completed — Other reasons | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse event unrelated to study drug | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 2 | 0 | 2 | 1 | 3 | 2
Not completed — Disease progression | 6 | 8 | 5 | 1 | 9 | 9 | 4 | 6 | 10 | 7 | 4 | 1 | 1 | 25 | 22 | 2 | 10 | 1 | 18 | 28
Not completed — Study drug toxicity | 0 | 1 | 4 | 0 | 1 | 2 | 4 | 2 | 2 | 0 | 6 | 1 | 2 | 19 | 19 | 0 | 18 | 3 | 11 | 7
Not completed — Participant request to discontinue study treatment | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Participant withdrew consent | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 4 | 2
Not completed — Randomized but not treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1A: BMS-986249 240 mg Monotherapy | Part 1A: BMS-986249 800 mg Monotherapy | Part 1A: BMS-986249 1600 mg Monotherapy | Part 1A: BMS-986249 2400 mg Monotherapy | Part 1A: BMS-986249 1600 mg Q8W Monotherapy | Part 1B: BMS-986249 240 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q4W+ Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q8W + Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q8W+ Nivolumab Combination | Part 1B: BMS-986249 1600 mg Q8W+ Nivolumab Combination | Part 2A: Melanoma Arm A: BMS-986249 240 mg Q3W + Nivolumab 360 mg Q3W | Part 2A: Melanoma Arm B: BMS-986249 800 mg + Nivolumab 480 mg Q4W | Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2A: Melanoma Arm D: Ipilimumab 3 mg/kg Q3W + Nivolumab 1 mg/kg Q3W | Part 2A: Melanoma Arm E: Nivolumab 480 mg Q4W Monotherapy | Part 2A: Melanoma Arm F: BMS-986249 600 mg Q4W + Nivolumab 480 mg Q4W | Part 2B: Cohort 1 (Advanced or Intermediate HCC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg IV Q4W | Part 2B: Cohort 2 (Metastatic CRPC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2B: Cohort 3 (Unresectable TNBC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Total
Number analyzed (Participants) | 6 | 11 | 10 | 1 | 11 | 12 | 11 | 9 | 13 | 9 | 10 | 3 | 3 | 58 | 59 | 3 | 36 | 5 | 41 | 45 | 356
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.0 (18.9) | 64.8 (7.5) | 60.4 (10.2) | 64 (NA) — Insufficient number of participants to calculate SD | 60.3 (11.6) | 56.3 (8.8) | 53.9 (12.4) | 61.4 (11.2) | 55.3 (11.4) | 59.0 (8.0) | 60.1 (9.9) | 60.7 (13.6) | 73.3 (7.6) | 61.4 (14.7) | 57.3 (13.8) | 59.7 (24.8) | 60.3 (12.4) | 60.4 (9.8) | 68.6 (8.0) | 51.2 (12.8) | 59.4 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 8 | 0 | 7 | 9 | 4 | 1 | 4 | 5 | 4 | 1 | 1 | 22 | 27 | 1 | 19 | 1 | 0 | 45 | 170
  Male | 3 | 3 | 2 | 1 | 4 | 3 | 7 | 8 | 9 | 4 | 6 | 2 | 2 | 36 | 32 | 2 | 17 | 4 | 41 | 0 | 186
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 1 | 2 | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 7 | 11 | 0 | 2 | 1 | 3 | 3 | 39
  Not Hispanic or Latino | 5 | 10 | 8 | 0 | 7 | 10 | 10 | 6 | 10 | 8 | 6 | 3 | 1 | 11 | 8 | 1 | 11 | 1 | 6 | 13 | 135
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 3 | 2 | 1 | 2 | 0 | 1 | 40 | 40 | 2 | 23 | 3 | 32 | 29 | 182
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 9
  White | 4 | 11 | 7 | 1 | 8 | 11 | 11 | 6 | 9 | 9 | 10 | 3 | 3 | 57 | 57 | 3 | 36 | 5 | 40 | 44 | 335
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) - Part 1 A and 1 B
Description: Adverse Events (AEs):
  Adverse events are any unwanted or harmful medical occurrences in a participant who receives a study drug or intervention. These events may or may not be related to the treatment.
  Serious Adverse Events (SAEs):
  Serious adverse events are adverse events that result in death, are life-threatening, require hospitalization or prolong existing hospitalization, cause significant disability or incapacity, or result in a birth defect.
Time Frame: From first dose until 100 days after last dose of study therapy (up to approximately 38 weeks)
Population: All treated participants in Part 1 A and B. Prespecified to be reported for Part 1 A and 1 B only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: BMS-986249 240 mg Monotherapy | Part 1A: BMS-986249 800 mg Monotherapy | Part 1A: BMS-986249 1600 mg Monotherapy | Part 1A: BMS-986249 2400 mg Monotherapy | Part 1A: BMS-986249 1600 mg Q8W Monotherapy | Part 1B: BMS-986249 240 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q4W+ Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q8W + Nivolumab Combination | Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 1B: BMS-986249 1600 mg Q8W+ Nivolumab Combination
Number analyzed (Participants) | 6 | 11 | 10 | 1 | 11 | 12 | 11 | 9 | 13 | 9 | 10
Participants
  Adverse events (AEs) | 6 | 11 | 10 | 1 | 11 | 12 | 11 | 9 | 13 | 9 | 10
  Serious adverse events (SAEs) | 4 | 8 | 8 | 1 | 7 | 8 | 7 | 7 | 10 | 7 | 8
  Adverse events (AEs) leading to discontinuation | 0 | 2 | 4 | 0 | 2 | 3 | 5 | 4 | 2 | 3 | 5

2. Primary Outcome: Number of Participants With Adverse Events (AEs) Meeting Protocol-Defined Dose-Limiting Toxicity (DLT) Criteria - Part 1 A and 1 B
Description: Dose-limiting toxicities (DLTs) were defined by the incidence, intensity, and duration of adverse events (AEs) possibly related to study treatment during the 5-week (35-day) DLT evaluation period for both BMS-986249 monotherapy and combination therapy. Participants who received at least 2 doses and completed or discontinued due to a DLT within this period were considered DLT-evaluable. Those who withdrew or received less than 2 doses for reasons other than a DLT were not DLT-evaluable and could be replaced. Any drug-related AE meeting DLT criteria resulted in discontinuation of study treatment. DLTs guided dose escalation and helped define the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D).
Time Frame: From first dose until 5 weeks after first dose of study medicine (up to approximately 5 weeks)
Population: All treated participants in Part 1 A and B who were evaluable for dose-limiting toxicities (DLT). Prespecified to be reported for Part 1 A and 1 B only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: BMS-986249 240 mg Monotherapy | Part 1A: BMS-986249 800 mg Monotherapy | Part 1A: BMS-986249 1600 mg Monotherapy | Part 1A: BMS-986249 2400 mg Monotherapy | Part 1A: BMS-986249 1600 mg Q8W Monotherapy | Part 1B: BMS-986249 240 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q4W+ Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q8W + Nivolumab Combination | Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 1B: BMS-986249 1600 mg Q8W+ Nivolumab Combination
Number analyzed (Participants) | 6 | 11 | 10 | 1 | 11 | 12 | 11 | 9 | 13 | 9 | 10
Participants | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3

3. Primary Outcome: Number of Participants Who Died - Part 1 A and 1 B
Description: Number of Participants who Died
Time Frame: From enrollment until the date of death from any cause (up to approximately 83 months)
Population: All treated participants in Part 1 A and B. Prespecified to be reported for Parts 1 A and 1 B only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: BMS-986249 240 mg Monotherapy | Part 1A: BMS-986249 800 mg Monotherapy | Part 1A: BMS-986249 1600 mg Monotherapy | Part 1A: BMS-986249 2400 mg Monotherapy | Part 1A: BMS-986249 1600 mg Q8W Monotherapy | Part 1B: BMS-986249 240 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q4W+ Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q8W + Nivolumab Combination | Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 1B: BMS-986249 1600 mg Q8W+ Nivolumab Combination
Number analyzed (Participants) | 6 | 11 | 10 | 1 | 11 | 12 | 11 | 9 | 13 | 9 | 10
Participants | 4 | 10 | 7 | 1 | 6 | 11 | 8 | 7 | 8 | 4 | 9

4. Primary Outcome: Number of Participants With Shifts From Baseline in Laboratory Tests Results - Part 1 A and 1 B
Description: Number of Participants with Shifts from Baseline in Laboratory Tests
Time Frame: From first dose until 100 days after last dose of study therapy (up to approximately 38 weeks)
Population: All treated participants in Part 1 A and B with baseline and post-baseline laboratory results. Prespecified to be reported for Parts 1 A and 1 B only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: BMS-986249 240 mg Monotherapy | Part 1A: BMS-986249 800 mg Monotherapy | Part 1A: BMS-986249 1600 mg Monotherapy | Part 1A: BMS-986249 2400 mg Monotherapy | Part 1A: BMS-986249 1600 mg Q8W Monotherapy | Part 1B: BMS-986249 240 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q4W+ Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q8W + Nivolumab Combination | Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 1B: BMS-986249 1600 mg Q8W+ Nivolumab Combination
Number analyzed (Participants) | 6 | 11 | 9 | 1 | 11 | 12 | 11 | 9 | 13 | 9 | 10
Participants
  HEMOGLOBIN | 3 | 4 | 7 | 1 | 4 | 10 | 9 | 6 | 7 | 4 | 7
  PLATELET COUNT | 1 | 1 | 2 | 0 | 0 | 0 | 3 | 0 | 2 | 1 | 3
  LEUKOCYTES, LOCAL LAB | 1 | 0 | 1 | 0 | 2 | 3 | 4 | 0 | 2 | 1 | 3
  ABSOLUTE NEUTROPHIL COUNT DRV | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 0 | 1 | 2 | 2
  LYMPHOCYTES (ABSOLUTE): number analyzed (Participants) | 2 | 3 | 3 | 0 | 2 | 2 | 2 | 1 | 2 | 2 | 1
  LYMPHOCYTES (ABSOLUTE) | 2 | 1 | 3 |  | 0 | 0 | 1 | 0 | 2 | 2 | 0
  LYMPHOCYTES (ABSOLUTE), LOCAL LAB: number analyzed (Participants) | 5 | 10 | 8 | 1 | 9 | 11 | 10 | 9 | 10 | 7 | 10
  LYMPHOCYTES (ABSOLUTE), LOCAL LAB | 2 | 7 | 6 | 0 | 3 | 6 | 5 | 5 | 1 | 6 | 4
  CREATININE, LOCAL LAB | 0 | 4 | 1 | 0 | 1 | 1 | 1 | 1 | 3 | 2 | 5
  ALKALINE PHOSPHATASE (ALP) LOCAL LAB | 1 | 7 | 1 | 1 | 3 | 5 | 4 | 6 | 5 | 2 | 6
  ALANINE AMINOTRANSFERASE (ALT), LOCAL LAB | 2 | 4 | 2 | 0 | 2 | 4 | 4 | 4 | 5 | 3 | 4
  ASPARTATE AMINOTRANSFERASE (AST), LOCAL LAB | 2 | 7 | 3 | 1 | 3 | 4 | 6 | 4 | 5 | 3 | 5
  BILIRUBIN, TOTAL, LOCAL LAB | 2 | 1 | 1 | 1 | 1 | 1 | 5 | 2 | 4 | 3 | 2

5. Primary Outcome: Number of Participants With Treatment-Related Grade 3-5 Adverse Events (AEs) Within 24 Weeks - Part 2 A Arms C, D and F, and Part 2 B
Description: Adverse Events (AEs):
  Adverse events are any unwanted or harmful medical occurrences in a participant who receives a study drug or intervention. These events may or may not be related to the treatment.
  Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; no intervention needed.
  Grade 2: Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate activities.
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling.
  Grade 4: Life-threatening consequences; urgent intervention required. Grade 5: Death related to the adverse event.
Time Frame: From first dose until 24 weeks after first dose (up to approximately 24 weeks)
Population: All treated participants in Part 2 A Arms C, D and F, and Part 2 B. Prespecified to be reported for Part 2 A Arms C, D and F, and Part 2 B only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2A: Melanoma Arm D: Ipilimumab 3 mg/kg Q3W + Nivolumab 1 mg/kg Q3W | Part 2A: Melanoma Arm F: BMS-986249 600 mg Q4W + Nivolumab 480 mg Q4W | Part 2B: Cohort 1 (Advanced or Intermediate HCC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg IV Q4W | Part 2B: Cohort 2 (Metastatic CRPC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2B: Cohort 3 (Unresectable TNBC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W
Number analyzed (Participants) | 58 | 59 | 36 | 5 | 41 | 45
Participants | 24 | 18 | 14 | 4 | 13 | 11

6. Primary Outcome: Objective Response Rate (ORR) as Assessed by Investigator - Part 2 A Arm C and F
Description: Objective response rate (ORR) is defined as the percent of participants whose best overall response (BOR) is either complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1:
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must also have reduction in the short axis to <10mm.
  Partial Response (PR): At least a30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From randomization until progression or death from any cause (up to approximately 83 months)
Population: All randomized participants in Part 2 A Arm C and F. Prespecified to be reported for Part 2 A Arm C and F only.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2A: Melanoma Arm F: BMS-986249 600 mg Q4W + Nivolumab 480 mg Q4W
Number analyzed (Participants) | 58 | 36
Percentage of participants | 36.2 [24.0 to 49.9] | 52.8 [35.5 to 69.6]

7. Secondary Outcome: Time to Deterioration in Part 2A (Arm C, D and F)
Description: TTD in Global Health Status/QoL and Physical Functioning will be defined as the time from randomization until a clinically meaningful decline (i.e., reduction ≥10 points) from baseline in EORTC QLQ-C30 global health/quality of life subscale score and Physical Functioning Scale score.
Time Frame: Approximately up to 6 months
Population: All Randomized Participants in Part 2A (Arm C, D and F)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2A: Melanoma Arm D: Ipilimumab 3 mg/kg Q3W + Nivolumab 1 mg/kg Q3W | Part 2A: Melanoma Arm F: BMS-986249 600 mg Q4W + Nivolumab 480 mg Q4W
Number analyzed (Participants) | 58 | 59 | 36
Months | 3.52 [1.87 to 5.29] | 4.37 [1.51 to 5.78] | 2.79 [1.22 to 5.65]

8. Secondary Outcome: Safety Related Events in Part 2A (Arm C, D and F) and 2B
Description: as for outcome 1
Time Frame: From first dose until 100 days after last dose of study therapy (up to approximately 38 weeks)
Population: All Treated Participants in Part 2A (Arm C, D and F) and 2B
Measure: Number; unit: Template
Arm/Group | Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2A: Melanoma Arm D: Ipilimumab 3 mg/kg Q3W + Nivolumab 1 mg/kg Q3W | Part 2A: Melanoma Arm F: BMS-986249 600 mg Q4W + Nivolumab 480 mg Q4W | Part 2B: Cohort 1 (Advanced or Intermediate HCC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg IV Q4W | Part 2B: Cohort 2 (Metastatic CRPC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2B: Cohort 3 (Unresectable TNBC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W
Number analyzed (Participants) | 57 | 58 | 36 | 5 | 41 | 45
Template
  Adverse Events | 57 | 57 | 35 | 5 | 40 | 45
  Serious Adverse Events | 41 | 28 | 20 | 5 | 29 | 25
  AEs leading to discontinuation | 24 | 25 | 20 | 4 | 13 | 13
  Deaths | 27 | 24 | 10 | 4 | 26 | 28

9. Secondary Outcome: BOR of PSA and PCWG3 Response Rate in Part 2B Cohort 2
Description: Best Overall Response (BOR) is defined as the best response recorded from the start of randomization or first dosing date until the date of objectively documented PD based on RECIST v1.1 criteria or PCWG3 (for prostate cancer), or the date of ubsequent therapy (including tumordirected radiotherapy and tumor-directed surgery which are not for palliative purpose), whichever occurs first.
Time Frame: From first dose (Parts 1 A and B) or randomization (Part 2 B) progression or death from any cause (up to approximately 83 months)
Population: All Treated Participants in Part 2B Cohort 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2B: Cohort 2 (Metastatic CRPC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W
Number analyzed (Participants) | 41
Percentage of participants
  PSA Response Rate | 14.6 [5.6 to 29.2]
  PCWG3 Response Rate | 9.8 [2.7 to 23.1]

10. Secondary Outcome: Progression Free Survival
Description: Defined as the time between the date of randomization (Part 2A), or first dosing for Part 1 and supplemental analysis in Part 2A, and the date of first documented tumor progression, based on investigator assessments (per RECIST v1.1 criteria or PCWG3), or death due to any cause, whichever occurs first.
Time Frame: as for outcome 9
Population: All Treated Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1A: BMS-986249 240 mg Monotherapy | Part 1A: BMS-986249 800 mg Monotherapy | Part 1A: BMS-986249 1600 mg Monotherapy | Part 1A: BMS-986249 2400 mg Monotherapy | Part 1A: BMS-986249 1600 mg Q8W Monotherapy | Part 1B: BMS-986249 240 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q4W+ Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q8W + Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q8W+ Nivolumab Combination | Part 1B: BMS-986249 1600 mg Q8W+ Nivolumab Combination | Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2A: Melanoma Arm D: Ipilimumab 3 mg/kg Q3W + Nivolumab 1 mg/kg Q3W | Part 2A: Melanoma Arm F: BMS-986249 600 mg Q4W + Nivolumab 480 mg Q4W | Part 2B: Cohort 1 (Advanced or Intermediate HCC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg IV Q4W | Part 2B: Cohort 2 (Metastatic CRPC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2B: Cohort 3 (Unresectable TNBC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W
Number analyzed (Participants) | 6 | 11 | 10 | 1 | 11 | 12 | 11 | 9 | 13 | 9 | 10 | 58 | 59 | 36 | 5 | 41 | 45
Months | 1.74 [1.41 to NA] — Insufficient number of events to calculate via KM methodology | 1.77 [1.15 to 1.84] | 1.69 [0.53 to 3.25] | 3.55 [NA to NA] — Insufficient number of events to calculate via KM methodology | 1.68 [1.05 to NA] — Insufficient number of events to calculate via KM methodology | 2.33 [1.68 to 3.32] | 1.71 [0.85 to 14.23] | 3.32 [1.22 to 4.40] | 1.92 [0.59 to 7.13] | 1.91 [1.02 to NA] — Insufficient number of events to calculate via KM methodology | 4.35 [0.92 to 12.45] | 6.51 [4.90 to 12.52] | 4.73 [2.89 to 9.76] | 10.38 [6.74 to NA] — Insufficient number of events to calculate via KM methodology | 2.99 [1.77 to NA] — Insufficient number of events to calculate via KM methodology | 5.62 [3.68 to 8.28] | 3.35 [1.84 to 5.36]

11. Secondary Outcome: Duration of Response
Description: Defined as the time between the date of first documented response (CR or PR) to the date of the first documented tumor progression, as determined by RECIST v1.1 or PCWG3 criteria, or death due to any cause, whichever occurs first. Subjects who start subsequent therapy without a prior reported progression will be censored at the last evaluable tumor assessments prior to initiation of the subsequent anticancer therapy. Subjects who die without a reported prior progression will be considered to have progressed on the date of their death. Subjects who neither progress nor die, DOR will be censored on the date of their last evaluable tumor assessment. DOR will be evaluated for responders (confirmed CR or PR) only.
Time Frame: as for outcome 9
Population: All Confirmed Responders
Measure: Median (Full Range); unit: Months
Arm/Group | Part 1A: BMS-986249 240 mg Monotherapy | Part 1A: BMS-986249 800 mg Monotherapy | Part 1A: BMS-986249 1600 mg Monotherapy | Part 1A: BMS-986249 2400 mg Monotherapy | Part 1A: BMS-986249 1600 mg Q8W Monotherapy | Part 1B: BMS-986249 240 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q4W+ Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q8W + Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q8W+ Nivolumab Combination | Part 1B: BMS-986249 1600 mg Q8W+ Nivolumab Combination | Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2A: Melanoma Arm D: Ipilimumab 3 mg/kg Q3W + Nivolumab 1 mg/kg Q3W | Part 2A: Melanoma Arm F: BMS-986249 600 mg Q4W + Nivolumab 480 mg Q4W | Part 2B: Cohort 1 (Advanced or Intermediate HCC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg IV Q4W | Part 2B: Cohort 2 (Metastatic CRPC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2B: Cohort 3 (Unresectable TNBC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 3 | 3 | 21 | 21 | 19 | 0 | 4 | 7
Months |  |  |  |  |  |  | NA [12.48 to NA] — Insufficient number of events to calculate via KM methodology |  | 15.80 [1.68 to NA] — Insufficient number of events to calculate via KM methodology | NA [1.74 to NA] — Insufficient number of events to calculate via KM methodology | NA [8.97 to NA] — Insufficient number of events to calculate via KM methodology | 26.84 [7.85 to NA] — Insufficient number of events to calculate via KM methodology | NA [7.2 to NA] — Insufficient number of events to calculate via KM methodology | NA [6.47 to NA] — Insufficient number of events to calculate via KM methodology |  | NA [NA to NA] — Insufficient number of events to calculate via KM methodology | 21.49 [3.68 to NA] — Insufficient number of events to calculate via KM methodology

12. Secondary Outcome: Time to Response
Description: Defined as the time from first dosing (Part 1)/randomization (Part 2A) to the date of the first confirmed documented response (CR or PR). TTR will be evaluated for responders (confirmed CR or PR) only.
Time Frame: From first dose to first objective response (Approximately up to 3 Months)
Population: All Confirmed Responders
Measure: Median (Full Range); unit: Months
Arm/Group | Part 1A: BMS-986249 240 mg Monotherapy | Part 1A: BMS-986249 800 mg Monotherapy | Part 1A: BMS-986249 1600 mg Monotherapy | Part 1A: BMS-986249 2400 mg Monotherapy | Part 1A: BMS-986249 1600 mg Q8W Monotherapy | Part 1B: BMS-986249 240 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q4W+ Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q8W + Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q8W+ Nivolumab Combination | Part 1B: BMS-986249 1600 mg Q8W+ Nivolumab Combination | Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2A: Melanoma Arm D: Ipilimumab 3 mg/kg Q3W + Nivolumab 1 mg/kg Q3W | Part 2A: Melanoma Arm F: BMS-986249 600 mg Q4W + Nivolumab 480 mg Q4W | Part 2B: Cohort 1 (Advanced or Intermediate HCC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg IV Q4W | Part 2B: Cohort 2 (Metastatic CRPC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2B: Cohort 3 (Unresectable TNBC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 3 | 3 | 21 | 21 | 19 | 0 | 4 | 7
Months |  |  |  |  |  |  | 2.76 [1.8 to 3.7] |  | 1.74 [1.7 to 3.9] | 3.48 [3.48 to 5.4] | 4.01 [3.5 to 4.3] | 2.86 [2.1 to 8.6] | 2.83 [2.0 to 26.4] | 2.83 [2.66 to 4.44] |  | 2.84 [1.7 to 3.9] | 1.87 [1.74 to 2.76]

13. Secondary Outcome: Objective Response Rate (ORR) as Assessed by Investigator - Part 1 A, 1B, 2A (Arms C,D,F) and 2B
Description: Objective response rate (ORR) is defined as the percent of participants whose best overall response (BOR) is either complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or Prostate Cancer Working Group (PCWG) 3. For both RECIST v1.1 and PCWG3:
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must also have reduction in the short axis to <10mm.
  Partial Response (PR): At least a30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: as for outcome 9
Population: All treated participants (Part 1A and B); all randomized participants (Part 2A and B).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1A: BMS-986249 240 mg Monotherapy | Part 1A: BMS-986249 800 mg Monotherapy | Part 1A: BMS-986249 1600 mg Monotherapy | Part 1A: BMS-986249 2400 mg Monotherapy | Part 1A: BMS-986249 1600 mg Q8W Monotherapy | Part 1B: BMS-986249 240 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q4W+ Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q8W + Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q8W+ Nivolumab Combination | Part 1B: BMS-986249 1600 mg Q8W+ Nivolumab Combination | Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2A: Melanoma Arm D: Ipilimumab 3 mg/kg Q3W + Nivolumab 1 mg/kg Q3W | Part 2A: Melanoma Arm F: BMS-986249 600 mg Q4W + Nivolumab 480 mg Q4W
Number analyzed (Participants) | 6 | 11 | 10 | 1 | 11 | 12 | 11 | 9 | 13 | 9 | 10 | 3 | 59 | 36
Percentage of participants | 0 [0.0 to 45.9] | 0 [0.0 to 28.5] | 0 [0.0 to 30.8] | 0 [0.0 to 97.5] | 0 [0.0 to 28.5] | 0 [0.0 to 26.5] | 18.2 [2.3 to 51.8] | 0 [0.0 to 33.6] | 23.1 [5.0 to 53.8] | 33.3 [7.5 to 70.1] | 30.0 [6.7 to 65.2] | 31.0 [19.5 to 44.5] | 27.1 [16.4 to 40.3] | 50.0 [32.9 to 67.1]

14. Secondary Outcome: Cmax and Ctau of BMS-986249 - Part 1 A and B, Part 2 A Arms C and F, Part 2 B
Description: Cmax: The highest concentration of BMS-986249 in the blood after dosing. Ctau: The concentration of BMS-986249 in the blood at the end of a dosing interval, just before the next dose
Time Frame: On Cycle 1 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1 (each cycle=28 days)
Population: All treated participants with baseline and at least one-post baseline PK result. Prespecified to be reported for Part 1 A and B, Part 2 A Arms C and F, Part 2 B only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1A: BMS-986249 240 mg Monotherapy | Part 1A: BMS-986249 800 mg Monotherapy | Part 1A: BMS-986249 1600 mg Monotherapy | Part 1A: BMS-986249 2400 mg Monotherapy | Part 1A: BMS-986249 1600 mg Q8W Monotherapy | Part 1B: BMS-986249 240 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q4W+ Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q8W + Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q8W+ Nivolumab Combination | Part 1B: BMS-986249 1600 mg Q8W+ Nivolumab Combination | Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2A: Melanoma Arm F: BMS-986249 600 mg Q4W + Nivolumab 480 mg Q4W | Part 2B: Cohort 1 (Advanced or Intermediate HCC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg IV Q4W | Part 2B: Cohort 2 (Metastatic CRPC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2B: Cohort 3 (Unresectable TNBC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W
Number analyzed (Participants) | 5 | 11 | 10 | 1 | 11 | 12 | 11 | 8 | 13 | 9 | 10 | 56 | 33 | 5 | 39 | 38
ng/mL
  Cmax Cycle 1 Day 1 | 398 (24) | 1451 (39) | 3569 (27) | 4965 (NA) — Insufficient number of participants with events to calculate | 2735 (31) | 454 (27) | 1322 (40) | 1729 (39) | 1397 (27) | 2105 (26) | 3146 (38) | 2274 (49) | 1114 (34) | 1752 (40) | 2050 (27) | 2404 (41)
  Cmax C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 3 | 3 | 0 | 0 | 0 | 0 | 0
  Cmax C3D1 |  |  |  |  | 2919 (48) |  |  |  | 1894 (33) | 1817 (32) | 2771 (28) |  |  |  |  |
  Cmax Cycle 4 Day 1: number analyzed (Participants) | 2 | 2 | 1 | 1 | 0 | 3 | 11 | 1 | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 0
  Cmax Cycle 4 Day 1 | 432 (55) | 1425 (14) | 5299 (NA) — Insufficient number of participants with events to calculate | 3910 (NA) — Insufficient number of participants with events to calculate |  | 570 (9) | 1706 (21) | 1436 (NA) — Insufficient number of participants with events to calculate |  |  |  |  | 930 (38) |  |  |
  Cmax C5D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0 | 0 | 0
  Cmax C5D1 |  |  |  |  |  |  |  |  |  |  |  | 2022 (50) |  |  |  |
  Ctau Cycle 1 Day 1: number analyzed (Participants) | 5 | 11 | 10 | 1 | 10 | 12 | 11 | 8 | 13 | 0 | 9 | 47 | 33 | 5 | 30 | 38
  Ctau Cycle 1 Day 1 | 7.69 (4151) | 174 (71) | 344 (418) | 385 (NA) — Insufficient number of participants with events to calculate | 52.6 (181) | 45.8 (322) | 143 (51) | 159 (58) | 20.2 (206) |  | 58.7 (190) | 57.9 (300) | 153 (34) | 82.3 (61) | 79.3 (98) | 66.2 (153)
  Ctau C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0
  Ctau C3D1 |  |  |  |  | 149 (24) |  |  |  | 94.4 (7) |  | 152 (45) |  |  |  |  |
  Ctau Cycle 4 Day 1: number analyzed (Participants) | 2 | 2 | 0 | 1 | 0 | 12 | 3 | 1 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0
  Ctau Cycle 4 Day 1 | 51.6 (255) | 1425 (14) |  | 236 (NA) — Insufficient number of participants with events to calculate |  | 170 (11) | 115 (310) | 107 (NA) — Insufficient number of participants with events to calculate |  |  |  |  | 151 (53) |  |  |
  CTau C5D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 0
  CTau C5D1 |  |  |  |  |  |  |  |  |  |  |  | 100 (83) |  |  |  |

15. Secondary Outcome: AUC(0-T) and AUC(TAU) of BMS-986249 - Part 1 A and B, Part 2 A Arms C and F, Part 2 B
Description: AUC(0-T): The total amount of BMS-986249 in the blood from the time it is given until a specific time point.
  AUC(TAU): The total amount of BMS-986249 in the blood over one dosing interval
Time Frame: On Cycle 1 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1 (each cycle=28 days)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part 1A: BMS-986249 240 mg Monotherapy | Part 1A: BMS-986249 800 mg Monotherapy | Part 1A: BMS-986249 1600 mg Monotherapy | Part 1A: BMS-986249 2400 mg Monotherapy | Part 1A: BMS-986249 1600 mg Q8W Monotherapy | Part 1B: BMS-986249 240 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q4W+ Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q8W + Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q8W+ Nivolumab Combination | Part 1B: BMS-986249 1600 mg Q8W+ Nivolumab Combination | Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2A: Melanoma Arm F: BMS-986249 600 mg Q4W + Nivolumab 480 mg Q4W | Part 2B: Cohort 1 (Advanced or Intermediate HCC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg IV Q4W | Part 2B: Cohort 2 (Metastatic CRPC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2B: Cohort 3 (Unresectable TNBC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W
Number analyzed (Participants) | 5 | 11 | 10 | 1 | 11 | 12 | 11 | 8 | 13 | 9 | 10 | 56 | 33 | 5 | 39 | 38
ng*h/mL
  AUC (0-T) Cycle 1 Day 1: number analyzed (Participants) | 5 | 11 | 10 | 1 | 10 | 12 | 11 | 8 | 13 | 9 | 9 | 47 | 31 | 5 | 30 | 38
  AUC (0-T) Cycle 1 Day 1 | 77826 (48) | 294432 (39) | 745654 (40) | 991294 (NA) — Insufficient number of participants with events to calculate | 671019 (48) | 96709 (49) | 292555 (32) | 378115 (31) | 325275 (35) | 521156 (36) | 688556 (29) | 612513 (44) | 255384 (23) | 653770 (7) | 638435 (24) | 696815 (34)
  AUC (Tau) Cycle 1 Day 1 | 67094 (53) | 288621 (37) | 629431 (55) | 999415 (NA) — Insufficient number of participants with events to calculate | 484593 (74) | 88780 (61) | 282516 (32) | 326037 (40) | 259533 (35) | 458972 (41) | 532540 (43) | 464205 (81) | 231346 (48) | 407104 (56) | 438370 (70) | 554691 (52)
  AUC (0-T) Cycle 4 Day 1: number analyzed (Participants) | 2 | 2 | 0 | 1 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0
  AUC (0-T) Cycle 4 Day 1 | 432 (55) | 284353 (45) |  | 687899 (NA) — Insufficient number of participants with events to calculate |  | 181278 (9) | 338096 (49) | 255093 (NA) — Insufficient number of participants with events to calculate |  |  |  |  | 260319 (35) |  |  |
  AUC (Tau) Cycle 4 Day 1: number analyzed (Participants) | 2 | 2 | 1 | 1 | 0 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 0
  AUC (Tau) Cycle 4 Day 1 | 51.6 (255) | 147763 (25) | 114154 (NA) — Insufficient number of participants with events to calculate | 536764 (NA) — Insufficient number of participants with events to calculate |  | 139951 (71) | 223315 (64) | 255093 (NA) — Insufficient number of participants with events to calculate |  |  |  |  | 229430 (37) |  |  |
  AUC (0-T) C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 3 | 3 | 0 | 0 | 0 | 0 | 0
  AUC (0-T) C3D1 |  |  |  |  | 1121470 (53) |  |  |  | 611831 (19) | 780896 (45) | 972214 (28) |  |  |  |  |
  AUC (Tau) C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 3 | 3 | 0 | 0 | 0 | 0 | 0
  AUC (Tau) C3D1 |  |  |  |  | 1121470 (53) |  |  |  | 611831 (19) | 780896 (45) | 937806 (25) |  |  |  |  |
  AUC (0-T) C5D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 0
  AUC (0-T) C5D1 |  |  |  |  |  |  |  |  |  |  |  | 675816 (33) |  |  |  |
  AUC (Tau) C5D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0 | 0 | 0
  AUC (Tau) C5D1 |  |  |  |  |  |  |  |  |  |  |  | 564180 (52) |  |  |  |

16. Secondary Outcome: Accumulation Index for Cmax (AI_Cmax) and Accumulation Index for AUC (AI_AUC) of BMS-986249 - Part 1 A and B, Part 2 A Arms C, D and F, Part 2 B
Description: AI_Cmax: How much the highest concentration of BMS-986249 increases after multiple doses compared to a single dose.
  AI_AUC: How much the total exposure to BMS-986249 increases after multiple doses compared to a single dose.
Time Frame: On Cycle 1 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1 (each cycle=28 days)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part 1A: BMS-986249 240 mg Monotherapy | Part 1A: BMS-986249 800 mg Monotherapy | Part 1A: BMS-986249 1600 mg Monotherapy | Part 1A: BMS-986249 2400 mg Monotherapy | Part 1A: BMS-986249 1600 mg Q8W Monotherapy | Part 1B: BMS-986249 240 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q4W+ Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800 mg Q8W + Nivolumab Combination | Part 1B: BMS-986249 1200 mg Q8W+ Nivolumab Combination | Part 1B: BMS-986249 1600 mg Q8W+ Nivolumab Combination | Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2A: Melanoma Arm F: BMS-986249 600 mg Q4W + Nivolumab 480 mg Q4W | Part 2B: Cohort 1 (Advanced or Intermediate HCC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg IV Q4W | Part 2B: Cohort 2 (Metastatic CRPC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W | Part 2B: Cohort 3 (Unresectable TNBC): BMS-986249 1200 mg Q8W + Nivolumab 480 mg Q4W
Number analyzed (Participants) | 5 | 11 | 10 | 1 | 11 | 12 | 11 | 8 | 13 | 9 | 10 | 56 | 33 | 5 | 39 | 38
ratio
  AI (AUC) Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AI Cmax Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AI (AUC) Cycle 4 Day 1: number analyzed (Participants) | 2 | 2 | 0 | 1 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0
  AI (AUC) Cycle 4 Day 1 | 1.29 (11) | 1.07 (29) |  | 0.694 (NA) — Insufficient number of participants with events to calculate |  | 1.54 (1) | 1.23 (16) | 1.29 (NA) — Insufficient number of participants with events to calculate |  |  |  |  | 0.971 (24) |  |  |
  AI Cmax Cycle 4 Day 1: number analyzed (Participants) | 2 | 1 | 1 | 1 | 0 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 0
  AI Cmax Cycle 4 Day 1 | 1.02 (14) | 324 (NA) — Insufficient number of participants with events to calculate | 1.32 (NA) — Insufficient number of participants with events to calculate | 0.788 (NA) — Insufficient number of participants with events to calculate |  | 1.28 (10) | 1.25 (17) | 1.62 (NA) — Insufficient number of participants with events to calculate |  |  |  |  | 0.899 (64) |  |  |
  AI (AUC) C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 3 | 3 | 0 | 0 | 0 | 0 | 0
  AI (AUC) C3D1 |  |  |  |  | 1.35 (7) |  |  |  | 1.82 (43) | 1.3 (17) | 1.46 (11) |  |  |  |  |
  AI Cmax C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 3 | 3 | 0 | 0 | 0 | 0 | 0
  AI Cmax C3D1 |  |  |  |  | 1.17 (3) |  |  |  | 1.58 (85) | 0.918 (16) | 0.978 (14) |  |  |  |  |
  AI (AUC) C5D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 0 | 0 | 0 | 0
  AI (AUC) C5D1 |  |  |  |  |  |  |  |  |  |  |  | 1.13 (18) |  |  |  |
  AI Cmax C5D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 0 | 0 | 0 | 0
  AI Cmax C5D1 |  |  |  |  |  |  |  |  |  |  |  | 1.11 (53) |  |  |  |

17. Secondary Outcome: Number of Participants With Shifts From Baseline in Laboratory Test Results - Part 2A (Arms C and F) and 2B
Description: Number of Participants with Shifts from Baseline in Laboratory Tests
Time Frame: From first dose until 100 days after last dose of study therapy (up to approximately 38 weeks)
Population: All treated participants in Part 2A (Arms C,D, F) and B with baseline and post-baseline laboratory results. Prespecified to be reported for Parts 2A (Arms C,D,F) and 2B only.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q6W + Nivolumab 480 mg Q4W; Part 2A: Melanoma Arm F: BMS-986249 1200 mg Q6W + Nivolumab 480 mg Q4W; Part 2B: Cohort 1 (Advanced or Intermediate HCC):; Part 2B: Cohort 2 (Metastatic CRPC): BMS-986249 1200 mg Q6W + Nivolumab 480 mg Q4W; Part 2B: Cohort 3 (Unresectable TNBC): BMS-986249 1200 mg Q6W + Nivolumab 480 mg Q4W: BMS-986249 1200 mg IV every 6 weeks (Q6W) + nivolumab 480 mg IV every 4 weeks (Q4W), up to 2 years.
- Part 2A: Melanoma Arm D: Ipilimumab 3 mg/kg Q3W + Nivolumab 1 mg/kg Q3W: Ipilimumab 3 mg/kg IV every 3 weeks (Q3W) + nivolumab 1 mg/kg IV Q3W (4 doses), then nivolumab 480 mg IV every 4 weeks (Q4W), monotherapy, up to 2 years.
Arm/Group | Part 2A: Melanoma Arm C: BMS-986249 1200 mg Q6W + Nivolumab 480 mg Q4W | Part 2A: Melanoma Arm D: Ipilimumab 3 mg/kg Q3W + Nivolumab 1 mg/kg Q3W | Part 2A: Melanoma Arm F: BMS-986249 1200 mg Q6W + Nivolumab 480 mg Q4W | Part 2B: Cohort 1 (Advanced or Intermediate HCC): | Part 2B: Cohort 2 (Metastatic CRPC): BMS-986249 1200 mg Q6W + Nivolumab 480 mg Q4W | Part 2B: Cohort 3 (Unresectable TNBC): BMS-986249 1200 mg Q6W + Nivolumab 480 mg Q4W
Number analyzed (Participants) | 57 | 58 | 36 | 5 | 41 | 45
Participants
  HEMOGLOBIN | 42 | 43 | 25 | 3 | 32 | 33
  PLATELET COUNT | 13 | 10 | 7 | 2 | 15 | 12
  LEUKOCYTES, LOCAL LAB | 12 | 10 | 6 | 0 | 9 | 14
  ABSOLUTE NEUTROPHIL COUNT DRV | 7 | 8 | 6 | 0 | 9 | 10
  LYMPHOCYTES (ABSOLUTE) | 9 | 19 | 10 | 0 | 11 | 11
  LYMPHOCYTES (ABSOLUTE), LOCAL LAB | 23 | 12 | 10 | 2 | 9 | 17
  CREATININE, LOCAL LAB | 20 | 17 | 10 | 3 | 14 | 5
  ALKALINE PHOSPHATASE (ALP) LOCAL LAB | 24 | 30 | 19 | 3 | 17 | 25
  ALANINE AMINOTRANSFERASE (ALT), LOCAL LAB | 38 | 40 | 23 | 4 | 18 | 27
  ASPARTATE AMINOTRANSFERASE (AST), LOCAL LAB | 27 | 40 | 22 | 3 | 19 | 31
  BILIRUBIN, TOTAL, LOCAL LAB | 12 | 18 | 7 | 3 | 12 | 5

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events: (From first dose to last dose + 100 days): Approximately 38 weeks All-Cause mortality (From randomization to end of study): Approximately 83 Months
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- Part 1A: BMS-986249 240mg Monotherapy: BMS-986249 240 mg IV Q4W
- Part 1A: BMS-986249 800mg Monotherapy: BMS-986249 800 mg IV Q4W
- Part 1A: BMS-986249 1600mg Q4W Monotherapy: BMS-986249 1600 mg IV Q4W
- Part 1A: BMS-986249 2400mg Monotherapy: BMS-986249 2400 mg IV Q4W
- Part 1A: BMS-986249 1600mg Q8WMonotherapy: BMS-986249 1600 mg IV Q8W
- Part 1B: BMS-986249 240mg Q4W + Nivolumab Combination: BMS-986249 240 mg IV Q4W + Nivolumab 480 mg IV Q4W
- Part 1B: BMS-986249 800mg Q4W + Nivolumab Combination: BMS-986249 800 mg IV Q4W + Nivolumab 480 mg IV Q4W
- Part 1B: BMS-986249 1200mg Q4W + Nivolumab Combination: BMS-986249 1200 mg IV Q4W + Nivolumab 480 mg IV Q6W
- Part 1B: BMS-986249 800mg Q8W+ Nivolumab Combination: BMS-986249 800 mg IV Q8W + Nivolumab 480 mg IV Q8W
- Part 1B: BMS-986249 1200mg Q8W+ Nivolumab Combination; Part 2B: Cohort 1 (HCC); Part 2B: Cohort 2 (Metastatic CRPC); Part 2B: Cohort 3 (Unresectable TNBC): BMS-986249 1200 mg IV Q8W + Nivolumab 480 mg IV Q8W
- Part 1B: BMS-986249 1600mg Q8W+ Nivolumab Combination: BMS-986249 1600 mg IV Q8W + Nivolumab 480 mg IV Q4W
- Part 2A: Melanoma Arms BMS-986249 240mg IV Q3W: BMS-986249 240 mg IV Q3W + Nivolumab 360 mg IV Q3W (14 doses), then Nivolumab 480 mg IV Q4W (maintenance)
- Part 2A: Melanoma Arms BMS-986249 800mg IV Q3W: BMS-986249 800 mg IV Q3W + Nivolumab 480 mg IV Q3W (14 doses), then Nivolumab 480 mg IV Q4W (maintenance)
- Part 2A: Melanoma Arms BMS-986249 1200mg IV Q3W: BMS-986249 1200 mg IV Q3W + Nivolumab 480 mg IV Q3W (14 doses), then Nivolumab 480 mg IV Q4W (maintenance)
- Part 2A: Melanoma Arms Ipilimumab 3mg/kg IV Q3W: Ipilimumab 3 mg/kg IV Q3W + Nivolumab 1 mg/kg IV Q3W (4 doses), then Nivolumab 480 mg IV Q4W (maintenance), up to 2 years
- Part 2A: Melanoma Arms Nivolumab Mono: Nivolumab 480 mg IV Q4W Monotherapy
- Part 2A: Melanoma Arms BMS-986249 600mg IV Q8W: BMS-986249 600 mg IV Q8W + Nivolumab 480 mg IV Q8W (Melanoma-specific combination)
Arm/Group | Part 1A: BMS-986249 240mg Monotherapy | Part 1A: BMS-986249 800mg Monotherapy | Part 1A: BMS-986249 1600mg Q4W Monotherapy | Part 1A: BMS-986249 2400mg Monotherapy | Part 1A: BMS-986249 1600mg Q8WMonotherapy | Part 1B: BMS-986249 240mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 1200mg Q4W + Nivolumab Combination | Part 1B: BMS-986249 800mg Q8W+ Nivolumab Combination | Part 1B: BMS-986249 1200mg Q8W+ Nivolumab Combination | Part 1B: BMS-986249 1600mg Q8W+ Nivolumab Combination | Part 2A: Melanoma Arms BMS-986249 240mg IV Q3W | Part 2A: Melanoma Arms BMS-986249 800mg IV Q3W | Part 2A: Melanoma Arms BMS-986249 1200mg IV Q3W | Part 2A: Melanoma Arms Ipilimumab 3mg/kg IV Q3W | Part 2A: Melanoma Arms Nivolumab Mono | Part 2A: Melanoma Arms BMS-986249 600mg IV Q8W | Part 2B: Cohort 1 (HCC) | Part 2B: Cohort 2 (Metastatic CRPC) | Part 2B: Cohort 3 (Unresectable TNBC)
All-Cause Mortality (participants affected / at risk) | 4/6 | 10/11 | 7/10 | 1/1 | 6/11 | 11/12 | 8/11 | 7/9 | 8/13 | 4/9 | 9/10 | 0/3 | 2/3 | 29/57 | 24/58 | 1/3 | 11/36 | 4/5 | 26/41 | 28/45
Serious Adverse Events (participants affected / at risk) | 4/6 | 8/11 | 8/10 | 1/1 | 7/11 | 8/12 | 7/11 | 7/9 | 10/13 | 7/9 | 8/10 | 3/3 | 1/3 | 42/57 | 28/58 | 1/3 | 20/36 | 5/5 | 29/41 | 25/45
Other Adverse Events (participants affected / at risk) | 6/6 | 11/11 | 9/10 | 1/1 | 9/11 | 12/12 | 11/11 | 9/9 | 12/13 | 9/9 | 10/10 | 3/3 | 3/3 | 57/57 | 57/58 | 3/3 | 34/36 | 5/5 | 39/41 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A: BMS-986249 240mg Monotherapy (N=6) | Part 1A: BMS-986249 800mg Monotherapy (N=11) | Part 1A: BMS-986249 1600mg Q4W Monotherapy (N=10) | Part 1A: BMS-986249 2400mg Monotherapy (N=1) | Part 1A: BMS-986249 1600mg Q8WMonotherapy (N=11) | Part 1B: BMS-986249 240mg Q4W + Nivolumab Combination (N=12) | Part 1B: BMS-986249 800mg Q4W + Nivolumab Combination (N=11) | Part 1B: BMS-986249 1200mg Q4W + Nivolumab Combination (N=9) | Part 1B: BMS-986249 800mg Q8W+ Nivolumab Combination (N=13) | Part 1B: BMS-986249 1200mg Q8W+ Nivolumab Combination (N=9) | Part 1B: BMS-986249 1600mg Q8W+ Nivolumab Combination (N=10) | Part 2A: Melanoma Arms BMS-986249 240mg IV Q3W (N=3) | Part 2A: Melanoma Arms BMS-986249 800mg IV Q3W (N=3) | Part 2A: Melanoma Arms BMS-986249 1200mg IV Q3W (N=57) | Part 2A: Melanoma Arms Ipilimumab 3mg/kg IV Q3W (N=58) | Part 2A: Melanoma Arms Nivolumab Mono (N=3) | Part 2A: Melanoma Arms BMS-986249 600mg IV Q8W (N=36) | Part 2B: Cohort 1 (HCC) (N=5) | Part 2B: Cohort 2 (Metastatic CRPC) (N=41) | Part 2B: Cohort 3 (Unresectable TNBC) (N=45)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Hypopituitarism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 2 | 1 | 0 | 2 | 0 | 0 | 2 | 2 | 2 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 3 | 0 | 4 | 0 | 0 | 2
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 2 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 1 | 0 | 2 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Immune-mediated hepatic disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Klebsiella urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Listeriosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 3
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 3 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6 | 1 | 1 | 1 | 3 | 4 | 5 | 3 | 2 | 2 | 0 | 0 | 6 | 6 | 1 | 3 | 1 | 4 | 2
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 1 | 4 | 5
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Immune-mediated nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bleeding varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A: BMS-986249 240mg Monotherapy (N=6) | Part 1A: BMS-986249 800mg Monotherapy (N=11) | Part 1A: BMS-986249 1600mg Q4W Monotherapy (N=10) | Part 1A: BMS-986249 2400mg Monotherapy (N=1) | Part 1A: BMS-986249 1600mg Q8WMonotherapy (N=11) | Part 1B: BMS-986249 240mg Q4W + Nivolumab Combination (N=12) | Part 1B: BMS-986249 800mg Q4W + Nivolumab Combination (N=11) | Part 1B: BMS-986249 1200mg Q4W + Nivolumab Combination (N=9) | Part 1B: BMS-986249 800mg Q8W+ Nivolumab Combination (N=13) | Part 1B: BMS-986249 1200mg Q8W+ Nivolumab Combination (N=9) | Part 1B: BMS-986249 1600mg Q8W+ Nivolumab Combination (N=10) | Part 2A: Melanoma Arms BMS-986249 240mg IV Q3W (N=3) | Part 2A: Melanoma Arms BMS-986249 800mg IV Q3W (N=3) | Part 2A: Melanoma Arms BMS-986249 1200mg IV Q3W (N=57) | Part 2A: Melanoma Arms Ipilimumab 3mg/kg IV Q3W (N=58) | Part 2A: Melanoma Arms Nivolumab Mono (N=3) | Part 2A: Melanoma Arms BMS-986249 600mg IV Q8W (N=36) | Part 2B: Cohort 1 (HCC) (N=5) | Part 2B: Cohort 2 (Metastatic CRPC) (N=41) | Part 2B: Cohort 3 (Unresectable TNBC) (N=45)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 3 | 0 | 1 | 6 | 1 | 3 | 5 | 1 | 4 | 1 | 2 | 27 | 31 | 2 | 13 | 1 | 21 | 23
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 4 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 1 | 0 | 0 | 2
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 6 | 2 | 0 | 2 | 0 | 5 | 2
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 1 | 0 | 0 | 9 | 12 | 1 | 1 | 1 | 5 | 4
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 3 | 1 | 0 | 0
Hypopituitarism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 4 | 2 | 1 | 1 | 0 | 13 | 12 | 0 | 8 | 1 | 4 | 8
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Eyelid irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Swelling of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 1 | 1 | 2 | 5 | 1 | 0 | 3 | 2 | 2 | 1 | 1 | 10 | 3 | 0 | 4 | 0 | 3 | 8
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 4 | 1 | 0 | 3
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 5 | 1 | 0 | 3 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 2 | 0 | 5 | 3 | 2 | 0 | 6 | 1 | 1 | 0 | 1 | 8 | 9 | 2 | 5 | 1 | 6 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 7 | 0 | 1 | 6 | 1 | 3 | 2 | 1 | 4 | 1 | 2 | 25 | 19 | 1 | 15 | 2 | 19 | 19
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 1 | 1 | 2
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 2 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 5 | 0 | 2 | 6 | 3 | 2 | 4 | 1 | 3 | 0 | 2 | 18 | 19 | 0 | 9 | 1 | 12 | 13
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 3
Vomiting (Gastrointestinal disorders) | 1 | 4 | 0 | 0 | 2 | 4 | 1 | 1 | 3 | 0 | 2 | 0 | 0 | 12 | 12 | 0 | 7 | 0 | 3 | 11
Application site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 13 | 5 | 1 | 3 | 0 | 3 | 7
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2
Complication associated with device (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related thrombosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 4 | 7 | 0 | 2 | 9 | 6 | 6 | 7 | 6 | 5 | 0 | 3 | 15 | 19 | 0 | 9 | 4 | 18 | 13
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hernia pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 2 | 0 | 0
Injection site extravasation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 0 | 2 | 0 | 2 | 3
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1 | 0 | 2 | 2 | 1 | 2 | 3 | 4 | 0 | 0 | 0 | 7 | 7 | 0 | 4 | 1 | 9 | 3
Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 0 | 0 | 5 | 4 | 3 | 4 | 1 | 1 | 1 | 1 | 14 | 11 | 0 | 8 | 3 | 3 | 14
Swelling face (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Xerosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 8 | 1 | 4 | 0 | 9 | 3
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 2 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 6 | 1 | 0 | 5 | 0 | 1 | 2
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 2
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 4 | 2 | 0 | 7 | 0 | 2 | 1
Campylobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 0
Norovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 5 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0
Spontaneous bacterial peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 6 | 0 | 3 | 1 | 6 | 8
Vascular access site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular access site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 2 | 3 | 2 | 1 | 0 | 2 | 25 | 22 | 1 | 14 | 2 | 10 | 16
Ammonia increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 2 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 9 | 7 | 2 | 6 | 0 | 1 | 10
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 1 | 1 | 1 | 2 | 1 | 2 | 1 | 3 | 2 | 0 | 2 | 21 | 25 | 0 | 10 | 2 | 8 | 17
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 6 | 0 | 1 | 0 | 4 | 7
Blood alkaline phosphatase increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 4 | 7 | 0 | 1 | 1 | 1 | 2
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 1 | 3 | 6 | 1 | 2 | 2 | 3 | 4
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 3 | 0 | 0 | 0 | 4 | 1
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 5 | 1 | 1 | 0 | 2 | 6
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 10 | 10 | 1 | 2 | 0 | 2 | 5
Blood creatinine increased (Investigations) | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 12 | 10 | 0 | 4 | 1 | 4 | 1
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 10 | 10 | 1 | 1 | 0 | 3 | 5
Blood lactic acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 9 | 0 | 2 | 0 | 2 | 10
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 0 | 3 | 1
Blood prolactin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 8 | 1 | 1 | 1 | 7 | 5
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 2
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 8 | 1 | 2 | 0 | 2 | 6
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 7 | 4 | 0 | 0 | 0 | 1 | 6
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 2 | 1 | 1 | 0 | 3 | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 11 | 13 | 1 | 7 | 0 | 5 | 8
Liver function test increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 2 | 5
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 1 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 5 | 0 | 1 | 0 | 4 | 2
Urine calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 2 | 5 | 0 | 8 | 0 | 13 | 5
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 4 | 0 | 2 | 3 | 5 | 1 | 4 | 1 | 3 | 0 | 0 | 10 | 17 | 0 | 7 | 1 | 16 | 13
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 4 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 3 | 2 | 0 | 4 | 0 | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 5 | 4 | 0 | 1 | 0 | 3 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 5 | 1 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 0 | 3 | 2 | 0 | 3 | 1 | 0 | 2 | 1 | 0 | 1 | 3 | 0 | 1 | 0 | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2 | 2 | 0 | 2 | 3 | 3 | 0 | 0 | 2 | 1 | 1 | 1 | 11 | 16 | 2 | 3 | 1 | 7 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 0 | 0 | 0 | 2 | 15 | 10 | 1 | 5 | 0 | 6 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 3 | 0 | 1 | 1 | 4 | 1 | 2 | 0 | 0 | 9 | 6 | 0 | 3 | 0 | 4 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 3 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 5 | 0 | 8 | 0 | 5 | 6
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 0 | 3 | 1 | 2 | 2
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 0 | 3 | 0 | 2 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 2 | 0 | 1 | 0 | 1 | 2
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 2 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 4 | 1 | 0 | 0 | 10 | 10 | 0 | 5 | 2 | 1 | 9
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 2
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 2 | 2 | 0 | 0 | 3 | 5 | 1 | 2 | 0 | 5 | 3
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 1 | 2 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 8 | 7 | 0 | 4 | 0 | 11 | 13
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 6 | 4 | 0 | 3 | 0 | 1 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 2 | 0 | 2 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 3 | 0 | 1 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acquired porokeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 1 | 0
Keloid scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukoplakia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 22 | 25 | 1 | 10 | 1 | 16 | 12
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 17 | 18 | 1 | 2 | 0 | 6 | 7
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 9 | 11 | 0 | 6 | 2 | 3 | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7 | 0 | 4 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 7 | 1 | 4 | 0 | 5 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 4 | 3 | 0 | 3 | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT03369223/Prot_SAP_000.pdf